CLINICAL TRIAL: NCT05079113
Title: Leveraging ctDNA Analysis to Improve Early Detection of Cancer Recurrence in the High-Risk Adjuvant Melanoma Setting
Brief Title: Leveraging ctDNA Analysis to Improve Early Detection of Cancer Recurrence in the High-Risk Melanoma Setting
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE1619
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Stage III Melanoma; Stage IV Cutaneous Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Retrospectively collected blood samples from a biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To generate meaningful data regarding ctDNA that would infer risk of recurrence in stage III melanoma patients.

DETAILED DESCRIPTION:
Cancer cells harbor and can acquire potentially hundreds of mutations, many of whom are found in the ctDNA. Circulating tumor DNA (ctDNA) holds the promise for the 50% of participants who do not need adjuvant therapies - participants could be monitored to ensure no increase in ctDNA. Participants treated could then be followed for the earliest possible blood level signs of recurrence (incr. ctDNA) and more quickly be switched to more effective therapies. Further, the treating physician could hold therapy until the first signs of ctDNA based recurrence for those participants that would benefit.

Blood sample from a biobank will be used to identify to monitor ctDNA. These blood samples were drawn at baseline, 3 months, 6 months and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Confirmed fully resected Stage IIIb-IV cutaneous melanoma; including patients treated neoadjuvantly within three months prior to resection.

Exclusion Criteria:

• Treatment plan inconsistent with the standard of care systemic adjuvant therapies 4.0 Study Design

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective biobanking samples collected at baseline, 3 months, 6 months and 18 months.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Identify a pattern for gene recognition of cancer recurrence earlier than standard of care. | samples taken at baseline, 3 months, 6 months and 18 months.
  Genomic sequencing of 40+ ctDNA genes will be analyzed to identify genetic alterations correlating with the development of recurrence in melanoma.

SECONDARY OUTCOMES:
Analyze the genetic pathway associated with cancer recurrence and biologic information. | samples taken at baseline, 3 months, 6 months and 18 months.
  The sequencing data will be analyzed against established determinants of cancer biology in clinically relevant melanoma variants identified via analysis of The Cancer Genome Atlas database.

CONTACTS AND LOCATIONS:
Overall Officials: James Isaacs, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer center, Cleveland, Ohio, United States